CLINICAL TRIAL: NCT01479998
Title: Novel Treatments to Enhance Smoking Cessation Before Cancer Surgery: Effects on Smoking and Surgical Outcomes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Reevaluating recruitment strategies
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1104008332; P50DA009241 (NIH)
Record Dates: First submitted 2011-11-04; First posted 2011-11-28 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; NRT nicotine replacement therapy; CBT cognitive behavioral therapy; contingency management
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care and nicotine replacement therapy (Active Comparator): standard care is 4 counseling sessions and nicotine replacement therapy
  Interventions: Other: standard care
- standard care plus NRT plus contingency management (Experimental): standard care is 4 counseling sessions and nicotine replacement therapy plus 3 weekly meetings with positive reinforcers
  Interventions: Other: standard care plus contingency management

INTERVENTIONS:
Other: standard care — standard care plus nicotine replacement therapy
  Arms: Standard care and nicotine replacement therapy
Other: standard care plus contingency management — standard care is 4 counseling sessions and nicotine replacement therapy plus 3 weekly meetings with positive reinforcers
  Arms: standard care plus NRT plus contingency management

SUMMARY:
Eligible participants will be randomized to either: 1) standard care (i.e., 4 counseling sessions and nicotine replacement therapy (NRT)) or 2) standard care + contingency management (i.e., 4 counseling sessions and NRT + 3x/week meetings with positive reinforcers)

DETAILED DESCRIPTION:
Participants will be recruited through the Thoracic Oncology Program and the Head and Neck Cancers Program. At the time of their initial surgical consultation, surgeons and their support staff in the Thoracic Oncology Program and Head and Neck Cancers Program will advise all of their patients about the present smoking cessation study as well as the Smoking Cessation Service at Smilow Cancer Hospital/Yale-New Haven Hospital and other resources in the community. Patients who express interest in the study and agree to quit smoking will be met at Smilow/YNHH for an intake appointment by a research assistant. Informed consent will be obtained prior to any other procedures, then during the intake session medical and tobacco use histories and breath carbon monoxide (CO) levels will be obtained from all participants. Study eligibility will be determined in concert with the surgeon and the principal investigator. As agreed upon by the surgeons, if participants meet eligibility criteria, their surgery will be scheduled for approximately 3 weeks after they enter the study.

Eligible participants will be randomized to either: 1) standard care (i.e., 4 counseling sessions and NRT) or 2) standard care + contingency management (i.e., 4 counseling sessions and NRT + 3x/week meetings with positive reinforcers). After this, all subjects will be met by a study therapist for their first counseling session, which is a preparation to quit session. The study counseling protocol will be based on practical counseling, which is a cognitive behavioral evidence based smoking cessation treatment modality (Fiore, Jaén et al. 2008). All participants will be asked to set a quit date within a week after this session. Consistent with the standard practice of the Smoking Cessation Service, all patients will receive pharmacotherapy in conjunction with counseling.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older,
2. smoking 5 or more cigarettes per day, and
3. diagnosed with any type of head, neck, or thoracic cancer,
4. agreement on a 3-week pre-surgical tobacco intervention by both patient and surgeon.

Exclusion Criteria:

1. Unstable psychiatric/medical conditions such as suicidal ideation, acute psychosis, severe alcohol dependence, or dementia,
2. history of allergic reactions to adhesives,
3. females of childbearing potential who are pregnant, nursing, or not practicing effective contraception.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
smoking cessation | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Toll, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Yale Cancer Center, New Haven, Connecticut